CLINICAL TRIAL: NCT05258929
Title: RElapse After Allograft: Link Between LoCus of Control and QualiTy of Life: REACT Study
Brief Title: RElapse After Allograft: Link Between LoCus of Control and QualiTy of Life
Acronym: REACT
Status: Terminated | Type: Observational
Why Stopped: low inclusion rate
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-1101; 2021-A02882-39 (Other: Agence Nationale de Sécurité des Médicaments et des produits de santé)
Record Dates: First submitted 2022-02-07; First posted 2022-02-28 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Allograft; Post-allograft Relapse
Keywords: hematology; allograft; relapse; psychological impact; locus of control
MeSH Terms: conditions — Recurrence | interventions — Data Collection; Lead; Transplantation, Homologous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hematological patients who underwent allograft: Patients who underwent allograft and then relapsed
  Interventions: Other: Data collection (Prior and planned treatments, allograft)

INTERVENTIONS:
Other: Data collection (Prior and planned treatments, allograft) — MHLC questionnaire (Multidimensional Health Locus of Control) when a novel therapeutic strategy is set up
  Other Names: Levenson Scale and QLQ-C30 at relapse

SUMMARY:
Allogeneic hematopoietic transplantation (AlloHCT) is a robust therapeutic that is used as a consolidation strategy in a number of haematological cancers. It provides durable responses as compared to chemotherapy alone. Despite the potential of the graft-versus-tumor effect that is driven by AlloHCT, relapse after AlloHCT remains common. Yet, the psychological impact of relapse after allograft is poorly appreciated.

DETAILED DESCRIPTION:
For patients with hematological cancers of poor prognosis (acute myeloid leukemia, myelodysplastic syndromes…), proceeding to allogeneic hematopoietic transplantation (AlloHCT) is the definitive curative approach. While AlloHCT is an invasive procedure, patients experience social isolation and distressing symptoms when hospitalized. Indeed, patients often report high levels of anxiety and/or depression during hospitalization and upon discharge. A number of risk factors have been linked to psychological morbidity and their impact on post-AlloHCT relapse have been less investigated. Of note, the health locus of control may play a significant role in determining patients' health-related behaviors. The health locus of control is defined as the set of beliefs a person has about his or her personal influence on health, including an internal locus of control (i.e. personal actions or thoughts can affect outcomes) and an external locus of control (i.e. outcome is believed to be determined by powerful others: God, health professionals, chance…). In this context, the aim of the study REACT is to identify the types of locus of control in relapsed patients after AlloHCT and the possible association with current disease perception as well as further therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Major patient who has been informed about the study;
* Allografted patient with molecular or clinical relapse.

Exclusion Criteria:

* Legal incapacity or limited capacity ; Medical or psychological incapacity or limited capacity;
* Not able to understand and complete surveys.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hematological patients who underwent allograft and are being diagnosed with relapse (molecular or clinical relapse)
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-04 (Actual); Study Completion 2022-06-04 (Actual)

PRIMARY OUTCOMES:
Correlation between the locus of control and the perception of the patient | 1 month
  Multidimensional Health Locus of Control questionnaire with regards to the locus of control. The survey contains 18-items with 6-items for each of its three subscales: Internal, Chance and Powerful Others. Each item is scored on a 6-point, Likert-type, scale from 1 (Strongly Disagree) to 6 (Strongly Agree). Scores for each subscale reflect the total score for the corresponding 6 items, with subscales having a minimum score of 6 and maximum score of 36.

SECONDARY OUTCOMES:
Correlation between the quality-of-life and the locus of control | 1 month
  QLQ-C30 questionnaire with regards to the locus of control. The maximum score is 126, the minimum score is 30. More the score is, worst the health state is.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Guyotat, PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No